CLINICAL TRIAL: NCT05111782
Title: Age Bias on Biopsychosocial Factors in Persons With Non-specific Low Back Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/1116 Aamer Naeem
Record Dates: First submitted 2021-10-07; First posted 2021-11-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will consist of persons with low back pain. This group will be further divided into groups for each decade.
  Interventions: Other: Symptom Modulation Approach, Movement Control Approach, Functional Optimization Approach
- Healthy Control Group (No Intervention): The control group will consist of healthy controls. This group will be further divided into groups for each decade.

INTERVENTIONS:
Other: Symptom Modulation Approach, Movement Control Approach, Functional Optimization Approach — Based on the patients' symptoms and level of disability, either symptom modulation or movement control or functional optimization exercises will be used. The exercises will be provided on alternate days for a duration of 30 minutes in each session preceded by electrotherapeutic modalities for pain relief and muscle relaxation. These modalities will be given for 15 min in each session. The total no. of sessions will be based on the patient's progress for a maximum of 4 weeks.
  Arms: Treatment Group

SUMMARY:
Low back pain is a debilitating condition experienced by people of all age groups. This study will be completed in two stages in which back pain assessment tools will be first translated to Urdu language and later on age-related bias on biopsychosocial factors will be assessed using various biopsychosocial tools over a period of six months.

DETAILED DESCRIPTION:
Low back pain (LBP) is an extremely common symptom experienced by people of all ages. The current incidence, prevalence and disability-adjusted life years (DALYs) account for 245.9 million cases/year (15th worldwide cause; 32.4% cases associated with leg pain), 577.0 million cases (15th worldwide cause) and 64.9 million DALYs (6th worldwide cause), respectively. In recent decades, the biopsychosocial model has been applied as a framework for understanding the complexity of low back pain disability in preference to a purely biomedical approach. Considering the large population of patients with LBP and limited medical resources, the development of brief and efficient prognostic clinical tools for use in routine practice is particularly significant. Recent data from epidemiological studies suggest that LBP could affect the physical function of young and older individuals differently. The age-related differ¬ences in the prevalence of some low back pathologies may explain the differential treatment outcomes. The aim of the study is to explore the age bias on biopsychosocial factors in persons with non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Both male & Female patients
2. Age group 20-60 Years
3. Diagnosed with nonspecific low back pain for more than 3 months (i.e., pain localized below the costal margin and above the inferior gluteal folds with or without referred leg pain of a nociceptive mechanical nature, not attributable to a recognizable, known specific spinal pathology, for a period of at least twelve weeks)

Exclusion Criteria:

Any serious conditions like neurological conditions which would not allow the patient to fill the questionnaire independently, any infection, tumor, spinal surgery, cognitive impairments, or any other rheumatologic disease would be excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 months
  The Numeric Pain Rating Scale will be used to quantify pain intensity on a scale of 1-10. A higher score represents higher pain.
Örebro Musculoskeletal Pain Screening Questionnaire | 6 months
  Screening for long term disability and failure to return to work will be done through Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ). The total score will range between 1 and 100. A higher score represents a poor outcome.
Keele STarT Back Screening Tool | 6 months
  Screening for primary care patients with low back pain to look for prognostic indicators that are relevant to initial decision making will be done through Keele STarT Back Screening Tool (SBST). Scores range from 0-9 and are produced by adding all positive items; patients who achieve a score of 0-3 are classified into the low-risk subgroup and those with scores of 4-9 into the medium-risk subgroup.
Low Back Outcome Scale | 6 months
  Pain & physical function will be assessed through the Low Back Outcome Scale. The Low Back Outcome Scale ranges from 0 to 75 and the higher score indicates better condition
Gait & Balance mobile Application | 6 months
  This mobile application will be used to measure the balance of the participants.
Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Sleep quality and disturbances will be assessed through Pittsburgh Sleep Quality Index (PSQI). The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The sub-scores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Center for Epidemiological Studies-Depression Scale (CES-D) | 6 months
  Depression symptoms will be evaluated through CES-D. The possible range is 0-60. If more than four questions are missing answers, do not score the CES-D questionnaire. A score of 16 points or more is considered depressed. The possible range is 0-60. A score of 16 points or more is considered depressed.
Fear Avoidance Belief Questionnaire (FABQ) | 6 months
  Fear of pain will be evaluated through FABQ. The score range is between 0 to 96. A higher score indicates strongly held fear-avoidance beliefs.
Job Content Questionnaire | 6 months
  Psychosocial aspects related to the job will be evaluated through the Job Content Questionnaire. The items are quantified on a four-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).
Roland Morris Disability Questionnaire (RMDQ) | 6 months
  Physical disability due to low back pain will be evaluated through RMDQ. The score can range from 0 to 24. A higher score indicates greater disability.
International Physical Activity Questionnaire (IPAQ) | 6 months
  Physical activity levels will be assessed through IPAQ. Data collected with IPAQ will be reported as a continuous measure and reported as median METminutes. walking is considered to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. A higher score indicates higher levels of physical activity.
Pain catastrophizing scale | 6 months
  Catastrophic thinking related to pain will be evaluated through the pain catastrophizing scale. It consists of 13 items scored from 0 to 4, resulting in a total possible score of 52. A higher score indicates a higher level of catastrophizing.
Pain self-efficacy Questionnaire (PSEQ) | 6 months
  Confidence in dealing with pain will be evaluated through PSEQ. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Force Platform | 6 months
  Standing postural control will be assessed using Force Platform.Coordinates of Centre of Pressure will be recorded.
Heart rate variability | 6 months
  Heart rate variability will be assessed through Smartwatch.
Sleep pattern | 6 months
  Sleep patterns will be assessed through Smartwatch in the form of phases of sleep and duration of sleep.
Activity level | 6 months
  Activity level will be assessed through Smartwatch in the form of the number of steps per day.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Foundation university institute of rehabilitation sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Hartvigsen J, Christensen K, Frederiksen H. Back pain remains a common symptom in old age. a population-based study of 4486 Danish twins aged 70-102. Eur Spine J. 2003 Oct;12(5):528-34. doi: 10.1007/s00586-003-0542-y. Epub 2003 May 14. PMID 12748896
- [Background] Urits I, Burshtein A, Sharma M, Testa L, Gold PA, Orhurhu V, Viswanath O, Jones MR, Sidransky MA, Spektor B, Kaye AD. Low Back Pain, a Comprehensive Review: Pathophysiology, Diagnosis, and Treatment. Curr Pain Headache Rep. 2019 Mar 11;23(3):23. doi: 10.1007/s11916-019-0757-1. PMID 30854609
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Hebert JJ, Koppenhaver SL, Walker BF. Subgrouping patients with low back pain: a treatment-based approach to classification. Sports Health. 2011 Nov;3(6):534-42. doi: 10.1177/1941738111415044. PMID 23016055
- [Background] Fritz JM, Brennan GP, Clifford SN, Hunter SJ, Thackeray A. An examination of the reliability of a classification algorithm for subgrouping patients with low back pain. Spine (Phila Pa 1976). 2006 Jan 1;31(1):77-82. doi: 10.1097/01.brs.0000193898.14803.8a. PMID 16395181